CLINICAL TRIAL: NCT04597567
Title: Clinical Outcome of Implant Removal Versus Retention After Posterior Fixation of Thoracolumbar Spine Fractures
Brief Title: Clinical Outcome of Implant Removal Versus Retention After Posterior Fixation of Thoracolumbar Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Samir Mondy, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Metal removal
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Thoracolumbar
Keywords: Metal removal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metal removal (Active Comparator)
  Interventions: Procedure: Metal removal
- Metal retention (No Intervention)

INTERVENTIONS:
Procedure: Metal removal — Implant removal after fracture consolidation after posterior fixation of thoracolumbar spine fractures
  Arms: Metal removal

SUMMARY:
Comparing clinical outcome between patients who underwent metal removal and those who retained the metal

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* Posterior fixation
* Six to nine months after fixation
* Neurologically free patient
* Fracture consolidation detected by ct
* Types A3&A4 fractures

Exclusion Criteria:

* unstable fractures B&C
* pathological fractures
* multilevel fractures
* poly trauma patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L questionnaire | Baseline
  Measuring the quality of life after metal removal

SECONDARY OUTCOMES:
Oswestry disability index | Baseline
  Measuring the quality of life after metal removal or without removal

REFERENCES:
- [Background] Court-Brown CM, Caesar B. Epidemiology of adult fractures: A review. Injury. 2006 Aug;37(8):691-7. doi: 10.1016/j.injury.2006.04.130. Epub 2006 Jun 30. PMID 16814787